CLINICAL TRIAL: NCT06041854
Title: Comparison Between Allograft and Enamel Matrix Derivative and Allograft in Treatment of Intrabony Defects
Brief Title: Allograft With Enamel Matrix Derivative Versus Allograft Alone in the Treatment of Intrabony Defects .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Rouida nouri, M.Sc. - Master Degree of Oral Medicine & Clinical Periodontology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02040122
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-03

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Intervention Model Description: Test group will receive EMD mixed with freeze-dried bone allograft, Control group will receive freeze-dried bone allograft
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- freeze-dried bone allograft combined with enamel matrix derivative (Experimental): The intrabony defects will be treated by surgical treatment and the defects filled by freeze-dried bone allograft mixed with enamel matrix derivative.
  Interventions: Procedure: Freeze-dried bone allograft combined with Enamel Matrix derivative
- freeze-dried bone allograft (Active Comparator): The intrabony defects will be treated by surgical treatment and the defects filled by freeze-dried bone allograft.
  Interventions: Procedure: Freeze-dried bone allograft

INTERVENTIONS:
Procedure: Freeze-dried bone allograft combined with Enamel Matrix derivative — The intrabony defects will be treated by minimally invasive surgical technique or modified minimally invasive surgical technique depending on defect extension, and the defects will be filled by freeze-dried bone allograft mixed with enamel matrix derivative.
  Enamel matrix derivatives are natural proteins that are produced in the developing dental follicle.The major components of EMD are amelogenins, a family of hydrophobic porcine tooth-derived proteins. They account for more than 95% of the total EMD protein content. Other proteins found in the enamel matrix include enamelin, ameloblastin, amelotin, apin and various proteinases, which have found in trace amounts in EMD. EMD adsorbs on decontamined root surfaces and alveolar bony defects and forms an insoluble scaffold complex.
  Arms: freeze-dried bone allograft combined with enamel matrix derivative
Procedure: Freeze-dried bone allograft — The intrabony defects will be treated by minimally invasive surgical technique or modified minimally invasive surgical technique depending on defect extension, and the defects will be filled by freeze-dried bone allograft .
  Allogeneic bone graft refers to bony tissue that is harvested from one individual and transplanted to a genetically different individual of the same species, principally osteoconductive, although it may have some osteoinductive capability, depending on how it is processed.
  Arms: freeze-dried bone allograft

SUMMARY:
Periodontal intrabony defects represent a major challenge for the clinician in periodontal therapy. If left untreated, these defects represent a risk factor for disease progression and additional attachment and bone loss.

All patients will receive full mouth scaling and root planing and be re-evaluated to assess patient cooperation and maintaining good oral hygiene. Subjects who showed persistent PPD ≥ 5 mm with radiographic evidence of periodontal intrabony defect presence will be included and will be randomly allocated to one of two treatment groups.One group will be treated by surgical treatment and the defects filled by freeze-dried bone allograft mixed with enamel matrix derivative. second group will be treated by surgical treatment and the defects filled by freeze-dried bone allograft .Clinical periodontal parameters (PI, GBI, PPD, CAL) will be re-evaluated at 3, 6 and 9 months after surgery. CBCT will be taken after 9 months of surgery and the defect measurements will be recorded

DETAILED DESCRIPTION:
primary goal of periodontal therapy is not arrest the tissue destruction caused periodontal disease only, but also to reconstruct the tissue lost caused by infectious process. Periodontal intrabony defects represent a major challenge for the clinician in periodontal therapy. If left untreated, these defects represent a risk factor for disease progression and additional attachment and bone loss. Surgical intervention is considered the treatment of choice for deep intrabony defects, which have not resolved following completion of cause-related periodontal therapy.

In general, periodontal studies showed that healing of periodontal defect after conventional periodontal therapy by collagenous tissue with epithelial cell migration within the gingival connective tissue and along the root surface. Therefore, a various of methods and techniques used to prevent epithelial ingrowth to the defect site and permit only a selective periodontal cells proliferation in attempt to regenerate periodontal tissues. Regenerative procedures including the use of certain types of bone replacement materials, barrier membranes, enamel matrix derivative (EMD), or various combinations thereof have been shown to facilitate periodontal regeneration characterized histologically by formation of root cementum, periodontal ligament, and alveolar bone and result superior in clinical, and radiographical patient reported outcomes compared to access flap surgery alone.

Various bone graft and bone substitutes materials can be helpful in the tissue restoration. This bone graft include autogenous bone graft, allografts, xenografts, and alloplastic materials. Autologous bone is considered the gold standard because of its biological activity due to vital cells and growth factors. Yet, the autologous bone from intra-oral donor sites is of restricted quantities and availability, and the bone tissue obtained from the iliac crest is described to show faster resorption. Moreover, the harvesting of autologous bone often requires a second surgical site associated with an additional bone defect, potential donor site morbidity limiting their application.

In recent years, the use of allogeneic human bone has been favored worldwide, and several histological and morphological studies have demonstrated that, there is no difference in the final stage of incorporation and new bone formation between allografts and autografts. Thus, the application of processed allogenic bone tissue is a reliable and predictable alternative.

Allogeneic bone graft refers to bony tissue that is harvested from one individual and transplanted to a genetically different individual of the same species, principally osteoconductive, although it may have some osteoinductive capability, depending on how it is processed.

Maxgraft® is allograft bone substitute processed by the Cells+Tissuebank Austria with a special cleaning process (Allotec® process). The purification process keeps the structural features and the interconnected macroporosity of human bone. It preserve natural bone structure and collagen content, therefore it serves as a scaffold for natural bone regeneration and has the potential of complete remodeling into patients' own bone. It is available as purely cancellous as well as cortico-cancellous granules and blocks.

Recently, better outcomes have been reported with a combination of xenograft and enamel matrix derivative (EMD) as it combines the osteoconductive and space-making properties of bone grafts with the ability of bioactive materials to stimulate periodontal regeneration. The major components of EMD are amelogenins, a family of hydrophobic porcine tooth-derived proteins. They account for more than 95% of the total EMD protein content. Other proteins found in the enamel matrix include enamelin, ameloblastin, amelotin, apin and various proteinases, which have found in trace amounts in EMD. EMD adsorbs on decontamined root surfaces and alveolar bony defects and forms an insoluble scaffold complex.

To the best of our knowledge, no previous studies have been performed for assessment of the efficacy of using emdogain with maxgraft.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 30-50 years.
* Patients with stage III periodontitis, will be diagnosed on the basis of probing pocket depth and clinical attachment loss.
* Presence of at least one or more radiographically detectable intrabony defect with clinical periodontal pocket depth (PPD) ≥5 mm, clinical attachment loss ≥5 mm, and radiographic depth of the intrabony defect ≥3 mm.
* No periodontal therapy within the last 6 months

Exclusion Criteria:

* Smoker and alcoholic patient.
* Patient with any signs, symptoms or history of systemic disease that might affect the periodontium and interfere with healing process.
* Pregnant patients.
* Patient who has traumatic occlusion.
* Uncooperative patient

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Radiographic bone defect fill | at baseline and 9 months
  Cone Beam Computed Tomography (CBCT) will be taken prior to periodontal surgery and after 9 months.
  The amount of reduction in the IBD measurements (defect resolution)

SECONDARY OUTCOMES:
Clinical attachment level | CAL will be measured at base line, 3, 6, 9 months postoperative
  CAL will be measured from the CEJ to the bottom of the gingival sulcus/periodontal pocket using UNC periodontal probe at six sites per tooth
Probing pocket depth | PD will be measured at base line, 3, 6, 9 months postoperative
  PD will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using UNC periodontal probe at six sites per tooth.
Plaque Index | PI will be measured at base line, 3, 6, 9 months postoperative
  Plaque index will be taken as an indicator for the patient oral hygiene.
Gingival Bleeding Index | GBI will be measured at base line, 3, 6, 9 months postoperative
  GBI will be measured according to Ainamo & Bay (1975)

CONTACTS AND LOCATIONS:
Overall Officials: Jilan Youssef, Professor, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kinane DF, Stathopoulou PG, Papapanou PN. Periodontal diseases. Nat Rev Dis Primers. 2017 Jun 22;3:17038. doi: 10.1038/nrdp.2017.38. PMID 28805207
- [Background] Garrett S. Periodontal regeneration around natural teeth. Ann Periodontol. 1996 Nov;1(1):621-66. doi: 10.1902/annals.1996.1.1.621. PMID 9118274
- [Background] Papapanou PN, Wennstrom JL. The angular bony defect as indicator of further alveolar bone loss. J Clin Periodontol. 1991 May;18(5):317-22. doi: 10.1111/j.1600-051x.1991.tb00435.x. PMID 2066446
- [Background] Reynolds MA, Kao RT, Camargo PM, Caton JG, Clem DS, Fiorellini JP, Geisinger ML, Mills MP, Nares S, Nevins ML. Periodontal regeneration - intrabony defects: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S105-7. doi: 10.1902/jop.2015.140378. Epub 2014 Oct 15. PMID 25315019
- [Background] Cortellini P, Tonetti MS. Clinical concepts for regenerative therapy in intrabony defects. Periodontol 2000. 2015 Jun;68(1):282-307. doi: 10.1111/prd.12048. PMID 25867990
- [Background] Sculean A, Nikolidakis D, Nikou G, Ivanovic A, Chapple IL, Stavropoulos A. Biomaterials for promoting periodontal regeneration in human intrabony defects: a systematic review. Periodontol 2000. 2015 Jun;68(1):182-216. doi: 10.1111/prd.12086. PMID 25867987
- [Background] Nibali L, Koidou VP, Nieri M, Barbato L, Pagliaro U, Cairo F. Regenerative surgery versus access flap for the treatment of intra-bony periodontal defects: A systematic review and meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:320-351. doi: 10.1111/jcpe.13237. PMID 31860134
- [Background] Mertens C, Decker C, Seeberger R, Hoffmann J, Sander A, Freier K. Early bone resorption after vertical bone augmentation--a comparison of calvarial and iliac grafts. Clin Oral Implants Res. 2013 Jul;24(7):820-5. doi: 10.1111/j.1600-0501.2012.02463.x. Epub 2012 Mar 27. PMID 22458589
- [Background] Palmer W, Crawford-Sykes A, Rose RE. Donor site morbidity following iliac crest bone graft. West Indian Med J. 2008 Nov;57(5):490-2. PMID 19565981
- [Background] Al-Abedalla K, Torres J, Cortes AR, Wu X, Nader SA, Daniel N, Tamimi F. Bone Augmented With Allograft Onlays for Implant Placement Could Be Comparable With Native Bone. J Oral Maxillofac Surg. 2015 Nov;73(11):2108-22. doi: 10.1016/j.joms.2015.06.151. Epub 2015 Jun 20. PMID 26126920
- [Background] Schlee M, Dehner JF, Baukloh K, Happe A, Seitz O, Sader R. Esthetic outcome of implant-based reconstructions in augmented bone: comparison of autologous and allogeneic bone block grafting with the pink esthetic score (PES). Head Face Med. 2014 May 28;10:21. doi: 10.1186/1746-160X-10-21. PMID 24885136
- [Background] Roberts TT, Rosenbaum AJ. Bone grafts, bone substitutes and orthobiologics: the bridge between basic science and clinical advancements in fracture healing. Organogenesis. 2012 Oct-Dec;8(4):114-24. doi: 10.4161/org.23306. Epub 2012 Oct 1. PMID 23247591
- [Background] Lorenz J, Schlee M, Al-Maawi S, Chia P, Sader RA, Ghanaati S. Variant Purification of an Allogeneic Bone Block. Acta Stomatol Croat. 2017 Jun;51(2):141-147. doi: 10.15644/asc51/2/7. PMID 28827851
- [Background] Trajkovski B, Jaunich M, Muller WD, Beuer F, Zafiropoulos GG, Houshmand A. Hydrophilicity, Viscoelastic, and Physicochemical Properties Variations in Dental Bone Grafting Substitutes. Materials (Basel). 2018 Jan 30;11(2):215. doi: 10.3390/ma11020215. PMID 29385747
- [Background] Corbella S, Alberti A, Calciolari E, Taschieri S, Francetti L. Enamel matrix derivative for the treatment of partially contained intrabony defects: 12-month results. Aust Dent J. 2019 Mar;64(1):27-34. doi: 10.1111/adj.12654. Epub 2018 Oct 15. PMID 30257036
- [Background] Lyngstadaas SP, Wohlfahrt JC, Brookes SJ, Paine ML, Snead ML, Reseland JE. Enamel matrix proteins; old molecules for new applications. Orthod Craniofac Res. 2009 Aug;12(3):243-53. doi: 10.1111/j.1601-6343.2009.01459.x. PMID 19627527
- [Background] Margolis HC, Beniash E, Fowler CE. Role of macromolecular assembly of enamel matrix proteins in enamel formation. J Dent Res. 2006 Sep;85(9):775-93. doi: 10.1177/154405910608500902. PMID 16931858
- [Background] Matarasso M, Iorio-Siciliano V, Blasi A, Ramaglia L, Salvi GE, Sculean A. Enamel matrix derivative and bone grafts for periodontal regeneration of intrabony defects. A systematic review and meta-analysis. Clin Oral Investig. 2015 Sep;19(7):1581-93. doi: 10.1007/s00784-015-1491-7. Epub 2015 May 27. PMID 26008887
- [Background] Lee MJ, Kim BO, Yu SJ. Clinical evaluation of a biphasic calcium phosphate grafting material in the treatment of human periodontal intrabony defects. J Periodontal Implant Sci. 2012 Aug;42(4):127-35. doi: 10.5051/jpis.2012.42.4.127. Epub 2012 Aug 31. PMID 22977742
- [Background] Cortellini P, Pini Prato G, Tonetti MS. Periodontal regeneration of human intrabony defects with titanium reinforced membranes. A controlled clinical trial. J Periodontol. 1995 Sep;66(9):797-803. doi: 10.1902/jop.1995.66.9.797. PMID 7500246
- [Background] Cornelini R, Scarano A, Piattelli M, Andreana S, Covani U, Quaranta A, Piattelli A. Effect of enamel matrix derivative (Emdogain) on bone defects in rabbit tibias. J Oral Implantol. 2004;30(2):69-73. doi: 10.1563/0.642.1. PMID 15119455
- [Background] Jung J, Park JS, Dard M, Al-Nawas B, Kwon YD. Effect of enamel matrix derivative liquid combined with synthetic bone substitute on bone regeneration in a rabbit calvarial model. Clin Oral Investig. 2021 Feb;25(2):547-554. doi: 10.1007/s00784-020-03473-4. Epub 2020 Aug 1. PMID 32740811